CLINICAL TRIAL: NCT06099626
Title: Study of Clinical Features and the Immune Mechanism Affecting Prognosis in Patients With Autoimmune Liver Disease Complicated With Covid-19 Infection
Brief Title: Study of Clinical Features of Patients With Autoimmune Liver Disease Complicated With Covid-19 and the Immune Mechanism Affecting Prognosis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023IITxG05
Record Dates: First submitted 2023-10-23; First posted 2023-10-25 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-08

CONDITIONS: Autoimmune Liver Disease, COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- A:autoimmune hepatitis
  Interventions: Other: Different types of disease
- B:autoimmune hepatitis/primary biliary cirrhosis
  Interventions: Other: Different types of disease
- C:/primary biliary cirrhosis
  Interventions: Other: Different types of disease
- D:Subjects tested positive for COVID-19 antigen or COVID-19 nucleic acid
  Interventions: Other: Different types of disease
- E: Subjects who have no previous history of COVID-19 infection and have been vaccinated against COVID-19.
  Interventions: Other: Different types of disease

INTERVENTIONS:
Other: Different types of disease — Groups were observed according to disease type

SUMMARY:
With the decreasing virulence of omicrons strain, the current domestic epidemic prevention policy has been changed based on the health of the people and the development needs of the country. At present, the infection rate of the novel coronavirus in China is rising rapidly. Previous studies have found that patients with chronic liver disease are more likely to be co-infected with coronavirus disease 2019 and have a worse prognosis. Based on its unique immune mechanism and therapeutic drugs, patients with autoimmune liver disease also have very different manifestations after infection with the novel coronavirus. By observing the clinical characteristics and prognosis of patients with autoimmune liver disease complicated with coronavirus disease 2019, this study analyzed the roles of vaccines, immunosuppressive agents and ursodeoxycholic acid , and explored the immune mechanism behind them, so as to seek new anti-coronavirus disease 2019 drugs and provide new strategies for clinical prevention and treatment.

ELIGIBILITY:
Group A: 1) Aged 18-75; 2) AIH patients diagnosed by AIH comprehensive scoring diagnosis system; 3) No history of other malignant tumors; 4) No metabolic diseases such as hypertension and diabetes; 5) No serious circulatory and respiratory diseases; 6) Non-alcoholic liver disease, drug-induced hepatitis, viral hepatitis and other liver diseases; 7) Exclude pregnant and lactating women.

Group B: 1) Aged 18-75 years; 2) Patients with PBC diagnosis; 3) No history of other malignant tumors; 4) No metabolic diseases such as hypertension and diabetes; 5) No serious circulatory and respiratory diseases; 6) Non-alcoholic liver disease, drug-induced hepatitis, viral hepatitis and other liver diseases; 7) Exclude pregnant and lactating women.

Group B: 1) Aged 18-75 years; 2) Patients with PBC diagnosis; 3) No history of other malignant tumors; 4) No metabolic diseases such as hypertension and diabetes; 5) No serious circulatory and respiratory diseases; 6) Non-alcoholic liver disease, drug-induced hepatitis, viral hepatitis and other liver diseases; 7) Exclude pregnant and lactating women.

Group B: 1) Aged 18-75 years; 2) Patients with PBC diagnosis; 3) No history of other malignant tumors; 4) No metabolic diseases such as hypertension and diabetes; 5) No serious circulatory and respiratory diseases; 6) Non-alcoholic liver disease, drug-induced hepatitis, viral hepatitis and other liver diseases; 7) Exclude pregnant and lactating women.

Group E: Those who had no previous history of COVID-19 infection and had been vaccinated against COVID-19.

-

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects were recruited from the Second Affiliated Hospital of Chongqing Medical University, and the postgraduate members/out-patient doctors/resident doctors of the research group were responsible for explaining the details of the study to the participants. After obtaining the written informed consent of the above subjects, the participants were included in the subject cohort (if the subjects had no corresponding understanding/behavioral ability, an agent would decide on their behalf). Some baseline data of patients were obtained by questionnaire. The number of participants included in this study refers to the number of participants included in the relevant literature.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Clinical features and prognosis | 6 months
  clinical manifestation,antibody titer

CONTACTS AND LOCATIONS:
Locations (1):
- Dazhi Zhang, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
The article is shared after publication